## Comparison of Ozone and Steroid Injection in Patients With Greater Trochanteric Pain Syndrome

## NCT04420572 - 01.03.2021

63 (sixty-three) patients were included in the study. Patients who were older than 18 years, had lateral hip pain for at least 3 months, had a VAS value of at least 4, had increased pain with pressing on the trochanter major, and failed conservative treatment were included in the study. The following patients were excluded from the study: Motor and/or sensory impairment compatible with radiculopathy, connective tissue disease, pregnancy, active infection, immune system disorders, untreated fracture, hip operation, steroid injection in the last 4 months, and/or hip region physical therapy, rheumatologic disease, cancer.

Evaluations were made before treatment (T0), 1 week after treatment (T1), and 1 month after treatment (T2). For the CSI group, T1 control was performed 1 week after CSI administration, and T2 control was performed 1 month after CSI administration. For the OI group, the T1 control was performed 1 week after the 4th OI administration, and the T2 control 1 month after the 4th OI administration. Physicians performing the administration and evaluation were different, thus allowing the study to be blinded. In the study, patients' Visual Analogue Scale (VAS), The Harris Hip Score (HHS) and The Nottingham Health Profile (NHP) questionnaires were filled. Patients were randomized into 2 groups according to Random Number Generation. The first group was determined as the ozone injection (OI) group and the second group as the corticosteroid injections (CSI) group.

33 patients were included in the 1st group and 30 patients in the 2nd group. The patients in the OI group received injections on the 1st, 4th, 7th and 10th days. A gas mixture containing 10 cc of 5% O3 and 95% medical O2 at a concentration of 25  $\mu$ g/ml in the first application, 20  $\mu$ g/ml in the second application, and 15  $\mu$ g/ml in the third and fourth applications was used. It was the same physician who prepared and administered ozone. Experience has shown that a single dose of ozone application is not sufficient, it must be applied in sessions for a strong effect. Therefore, we used 4 doses of OI instead of a single dose in our study. A single dose injection was given to the patients in the CSI group. The solution to be administered to the CSI group was obtained by mixing 1 ml of 2% lidocaine and 1 ml of betamethasone (Diprospan 2 mg/1ml+5 mg/1ml). It was the same physician who prepared and administered the solutions. In the studies, it was generally applied as a single dose and mixed with local anesthetic (LA). Therefore, in our study, we also applied it as a single dose by mixing it with LA. There will be pre-injection, postinjection 1st week and 1st month controls.